CLINICAL TRIAL: NCT03016000
Title: A Multicentre, Randomized Phase III Study of Thalidomide Maintenance Treatment in Patients With Diffuse Large B-cell Lymphoma
Brief Title: Thalidomide Maintenance Treatment in DLBCL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ru Feng, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFL2016-B2
Record Dates: First submitted 2016-11-02; First posted 2017-01-10 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: diffuse large B-cell lymphoma; Thalidomide; Maintenance
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Thalidomide; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thalidomide (Experimental): Thalidomide 50mg daily by mouth( increase 50mg after 2 weeks if tolerated until 200mg/day) until disease progression or intolerance due to AEs.The dose could be reduced if the patient experienced grade 2 or higher AEs. Does reductions for AEs were recommended (200 mg daily to 100 mg daily, 100 mg daily to 50 mg daily).In patients intolerant of 50mg/day, thalidomide discontinuation was allowed.
  Interventions: Drug: Thalidomide
- Observation (Other): Observation
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 50mg daily by mouth( increase 25mg after 2 weeks if tolerated Until 200mg/day) until disease progression or intolerance due to AEs.The dose could be reduced if patient experienced grade 2 or higher AEs. Does reductions for AEs were recommended (200 mg daily to 100 mg daily, 100 mg daily to 50 mg daily).In patients intolerant of 50mg/ day, thalidomide discontinuation was allowed.
  Other Names: Thalomid
  Arms: Thalidomide
Other: Observation — Just observation
  Arms: Observation

SUMMARY:
This is a randomized, multi-center,phase III study to evaluate the ability of thalidomide maintenance therapy to prolong relapse-free survival in diffuse large B cell lymphoma(DLBCL).

DETAILED DESCRIPTION:
This is a randomized, phase III study to evaluate the ability of thalidomide maintenance therapy to prolong relapse-free survival(RFS), in diffuse large B cell lymphoma(DLBCL).Patients will be enrolled after successful standard induction therapy (CR or CRu following standard R-CHOP-like therapy with 8 infusions of rituximab plus CHOP-like chemotherapy (4-8 cycles). Patients will be followed until an event occurs as defined in the protocol. To evaluate the clinical efficacy of thalidomide maintenance therapy as compared to observation in patients with DLBCL who have achieved a complete remission after appropriate first-line therapy, measured by RFS, 226 patients with DLCBL will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* NCCN-IPI>1,
* Known IPI, cell of origin and DHL at time of diagnosis,
* Negative pregnancy test,
* Men must agree not to father a child during the therapy,
* 6 to 8 cycles R-CHOP/like, total of 8 x Rituximab,
* CR, CRu

Exclusion Criteria:

* Transformed lymphoma,
* Secondary malignancy,
* HIV positive,
* Evidence of CNS involvement,
* Cardiac dysfunction (systolic ejection fraction <50%),
* Creatinine > 2.0 mg/dl

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | 5 years
  RFS was defined as the time between randomization and any documentation of relapse, death by any cause or last follow up.

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS was defined as the interval from randomization to death or the last follow-up for surviving patients.
Incidence of treatment-emergent adverse events | 5 years
  Adverse events were classified as defined by the National Cancer Institute Common Toxicity Criteria, version 2. Safety evaluations were focused especially on neurological symptoms and the development of deep venous thrombosis (DVT).

CONTACTS AND LOCATIONS:
Overall Officials: Ru Feng, M.D., Principal Investigator — Department of Hematology, Nanfang Hospital, Southern Medical University
Locations (1):
- Ru Feng, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chaganti S, Illidge T, Barrington S, Mckay P, Linton K, Cwynarski K, McMillan A, Davies A, Stern S, Peggs K; British Committee for Standards in Haematology. Guidelines for the management of diffuse large B-cell lymphoma. Br J Haematol. 2016 Jul;174(1):43-56. doi: 10.1111/bjh.14136. Epub 2016 May 16. No abstract available. PMID 27196701
- [Background] Michallet AS, Lebras L, Coiffier B. Maintenance therapy in diffuse large B-cell lymphoma. Curr Opin Oncol. 2012 Sep;24(5):461-5. doi: 10.1097/CCO.0b013e3283562036. PMID 22759738
- [Background] Aviles A, Cleto S, Huerta-Guzman J, Neri N. Interferon alfa 2b as maintenance therapy in poor risk diffuse large B-cell lymphoma in complete remission after intensive CHOP-BLEO regimens. Eur J Haematol. 2001 Feb;66(2):94-9. doi: 10.1034/j.1600-0609.2001.00272.x. PMID 11168516
- [Background] Gisselbrecht C, Schmitz N, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Milpied NJ, Radford J, Ketterer N, Shpilberg O, Duhrsen U, Hagberg H, Ma DD, Viardot A, Lowenthal R, Briere J, Salles G, Moskowitz CH, Glass B. Rituximab maintenance therapy after autologous stem-cell transplantation in patients with relapsed CD20(+) diffuse large B-cell lymphoma: final analysis of the collaborative trial in relapsed aggressive lymphoma. J Clin Oncol. 2012 Dec 20;30(36):4462-9. doi: 10.1200/JCO.2012.41.9416. Epub 2012 Oct 22. PMID 23091101
- [Background] Crump M, Leppa S, Fayad L, Lee JJ, Di Rocco A, Ogura M, Hagberg H, Schnell F, Rifkin R, Mackensen A, Offner F, Pinter-Brown L, Smith S, Tobinai K, Yeh SP, Hsi ED, Nguyen T, Shi P, Hahka-Kemppinen M, Thornton D, Lin B, Kahl B, Schmitz N, Savage KJ, Habermann T. Randomized, Double-Blind, Phase III Trial of Enzastaurin Versus Placebo in Patients Achieving Remission After First-Line Therapy for High-Risk Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2016 Jul 20;34(21):2484-92. doi: 10.1200/JCO.2015.65.7171. Epub 2016 May 23. PMID 27217449
- [Background] Witzens-Harig M, Benner A, McClanahan F, Klemmer J, Brandt J, Brants E, Rieger M, Meissner J, Hensel M, Neben K, Dreger P, Lengfelder E, Schmidt-Wolf I, Kramer A, Ho AD. Rituximab maintenance improves survival in male patients with diffuse large B-cell lymphoma. Results of the HD2002 prospective multicentre randomized phase III trial. Br J Haematol. 2015 Dec;171(5):710-9. doi: 10.1111/bjh.13652. Epub 2015 Oct 9. PMID 26449739
- [Background] Ji D, Li Q, Cao J, Guo Y, Lv F, Liu X, Wang B, Wang L, Luo Z, Chang J, Wu X, Hong X. Thalidomide enhanced the efficacy of CHOP chemotherapy in the treatment of diffuse large B cell lymphoma: A phase II study. Oncotarget. 2016 May 31;7(22):33331-9. doi: 10.18632/oncotarget.8973. PMID 27129176
- [Background] Maiolino A, Hungria VT, Garnica M, Oliveira-Duarte G, Oliveira LC, Mercante DR, Miranda EC, Quero AA, Peres AL, Barros JC, Tanaka P, Magalhaes RP, Rego EM, Lorand-Metze I, Lima CS, Renault IZ, Braggio E, Chiattone C, Nucci M, de Souza CA; Brazilian Multiple Myeloma Study Group (BMMSG/GEMOH). Thalidomide plus dexamethasone as a maintenance therapy after autologous hematopoietic stem cell transplantation improves progression-free survival in multiple myeloma. Am J Hematol. 2012 Oct;87(10):948-52. doi: 10.1002/ajh.23274. Epub 2012 Jun 23. PMID 22730113
- [Background] Spencer A, Prince HM, Roberts AW, Prosser IW, Bradstock KF, Coyle L, Gill DS, Horvath N, Reynolds J, Kennedy N. Consolidation therapy with low-dose thalidomide and prednisolone prolongs the survival of multiple myeloma patients undergoing a single autologous stem-cell transplantation procedure. J Clin Oncol. 2009 Apr 10;27(11):1788-93. doi: 10.1200/JCO.2008.18.8573. Epub 2009 Mar 9. PMID 19273705